CLINICAL TRIAL: NCT05038189
Title: Comparison of Spine Posture, Trunk Position Sense and Gait Characteristics Among Different Sub-types of Axial Spondyloarthritis Patients and Healthy Controls
Brief Title: Evaluation of Spine Posture, Trunk Position Sense and Gait in Axial Spondyloarthritis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Necmettin Erbakan University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, YASEMİN AKKUBAK, Research Assistant, Necmettin Erbakan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PhD_Yakkubak
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Non-radiographic Axial Spondyloarthritis; Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis,; Non-radiographic Axial Spondyloarthritis; Spine posture; Gait
MeSH Terms: conditions — Non-Radiographic Axial Spondyloarthritis; Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ankylosing Spondylitis (Experimental): Study group
  Interventions: Diagnostic Test: Gait parameters
- Non-radiographic Axial Spondyloarthritis (Experimental): Study group
  Interventions: Diagnostic Test: Spine posture
- Healthy individuals (Experimental): Control group
  Interventions: Diagnostic Test: Trunk position sense

INTERVENTIONS:
Diagnostic Test: Gait parameters — Trunk position sense as indicated by trunk reposition errors (TRE) and spine posture (thoracic and lumbar curvature) will be measured with a digital inclinometer. Gait analyses (cadence, stride length, swing phase duration, step duration and double stand duration) will be evaluated.
  Other Names: Trunk position sense; Spine posture
  Arms: Ankylosing Spondylitis
Diagnostic Test: Spine posture — Trunk position sense as indicated by trunk reposition errors (TRE) and spine posture (thoracic and lumbar curvature) will be measured with a digital inclinometer. Gait analyses (cadence, stride length, swing phase duration, step duration and double stand duration) will be evaluated.
  Other Names: Gait parameters; Trunk position sense
  Arms: Non-radiographic Axial Spondyloarthritis
Diagnostic Test: Trunk position sense — Trunk position sense as indicated by trunk reposition errors (TRE) and spine posture (thoracic and lumbar curvature) will be measured with a digital inclinometer. Gait analyses (cadence, stride length, swing phase duration, step duration and double stand duration) will be evaluated.
  Other Names: Gait parameters; Spine posture
  Arms: Healthy individuals

SUMMARY:
Axial Spondyloarthritis (Ax-SpA) are chronic systemic inflammatory rheumatological diseases characterized by axial skeletal involvement and enthesitis. Sacroiliitis is the most prominent sign of the disease. The International Society for the Evaluation of Spondyloarthritis created a new classification for Ax-SpA in 2009. According to this classification, Ax-SpA; It is divided into two groups as ankylosing spondylitis (AS) and non-radiographic axial spondyloarthritis (nr-axSpA).

With the emergence of the term nr-axSpA, studies have begun to compare AS and nr-axSpA in terms of genetic, epidemiological and clinical features, treatment needs and response to treatment.However, more studies are needed to better understand the clinical features and symptoms of nr-axSpA patients.

The aim of this study was to determine the clinical features of patients with nr-axSpA and AS; To evaluate spine posture, trunk position sense and gait parameters, and also to compare these results with healthy individuals.

DETAILED DESCRIPTION:
There are no studies comparing spine posture, trunk position sense and gait parameters in patients with nr-axSpA and AS. It is important to determine the changes that occur in nr-axSpA patients in the early period. At the same time, taking the necessary precautions and following these patients with the rehabilitation process can ensure that the radiographic development is delayed or not at all in the future.

Hypotheses:

H1: Trunk position sense is different from each other in individuals with Nr-axSpA and AS.

H2: Spatio-temporal features of gait are different in individuals with Nr-axSpA and AS.

H3: Plantar pressure distribution is different in individuals with Nr-axSpA and AS.

The Location of the Research: The research is carried out in Konya Necmettin Erbakan University Meram Faculty of Medicine, Rheumatology Department. After obtaining the permission of the ethics committee, official permission was obtained from Necmettin Erbakan University Meram Medical Faculty Hospital Chief Physician to conduct the study.

ELIGIBILITY:
Inclusion Criteria:

For AS and nr-axSpA;

* Diagnosed with AS and nr-axSpA by a rheumatologist according to ASAS criteria,
* Diagnosed with AS and nr-axSpA at least two years ago,
* Volunteer to participate in the study,
* Individuals between the ages of 18-65 will be included in the study.

For Healthy volunteers;

* Volunteer to participate in the study,
* Individuals between the ages of 18-65 will be included in the study.

Exclusion Criteria:

For AS and nr-axSpA;

* Having orthopedic problems in the lower extremity,
* Locomotor disorders (fractures and prostheses) and / or osteoporosis,
* Having a history of lower extremity and spine surgery,
* Having neurological and cognitive problems,
* Having vision and hearing problems,
* Regular exercise,
* Individuals with kyphosis above 50 degrees will be excluded from the study.

For Healthy volunteers;

* Having any musculoskeletal, neurological and rheumatological diseases,
* Having any condition (advanced respiratory or orthopedic problems, fracture, sprain or spine surgery) that will prevent the evaluation,
* Regular exercise,
* Individuals who do not agree to participate in the study will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Gait analyses | 6 months
  The spatiotemporal parameters of gait will be evaluated using the Diagnostic Support Baropodometer Footscan® 3D system. The spatial parameters of gait, step length (cm), step width (cm) and foot angle (degrees) and the temporal parameters of gait, speed (m/min), cadence (step/min) and stance time (sec) will be recorded. For evaluating of the plantar pressure distribution will be used the Diagnostic Support Baropodometer Footscan® 3D system, besides the dynamic evaluation and recording of the spatiotemporal parameters, the data on the total load on the forefoot, midfoot and hindfoot; the average pressure; and the distribution of load in the forefoot, midfoot and hindfoot will be also obtained.
Spine posture | 6 months
  Thoracic and lumbar curvature tests will be performed with a digital inclinometer (Acumar®, Dual Digital Inclinometer, Lafayette Instrument Company, IN, USA). For throcic curvature, the 7th cervical vertebra, the most prominent spinous process, and the sacrum will be used as reference points to palpate the spinal processes of T1-T2 and T12-L1, respectively. The feet of the inclinometers will be placed as simultaneously as possible over T1-T2 and T12-L1. The angle on the digital display of the inclinometer will be recorded as degree. The mean of three successful measurements will be used. For lumbar curvature, the sacrum and iliac crest will be used as reference points to palpate the spinal processes of T12-L1 and L5-S1, respectively. The feet of the inclinometers will be placed as simultaneously as possible over T12-L1 and L5-S1. The angle on the digital display of the inclinometer will be recorded in degrees.
Trunk position sense | 6 months
  Trunk position sense, as indicated by trunk reposition errors (TRE), will be assessed with a digital inclinometer (Acumar®,Dual Digital Inclinometer, Lafayette Instrument Company, IN, USA). The participants will be asked to stand upright in a comfortable position. The inferior angle of the scapula will first palpated as a bony landmark to find the spinousprocess of T4. After the placement of the inclinometer over the spinous process of T4, the participants will be asked to flex the trunk approximately 30° in the sagittal plane and hold this position for 3 s in eyes closed position. After returning to the neutral upright position, they will be asked to duplicate the previously attained position and held the position for 3 s for five times in a row. The absolute differences between the original position and the other five attempts will be recorded. The highest and lowest scores will be discarded and the mean of the tree remaining scores will be used to assess the trunk position sense.

SECONDARY OUTCOMES:
Stabilometric test | 6 months
  In the stabilometric evaluation, a STABYLO platform, which is produced by Diagnostic Support, will be used. A 40x80 cm sensing surface with 12,800 active sensors is used for the examination of body oscillations in the upright position (the foot at 30°) and for the evaluation of body strategies in a specific time frame (maximum 51.2 sec) by maintaining the eyes in the open and closed positions. In the present study, the body oscillations with open and closed eyes will be calculated as an area in cm².
Bath Ankylosing Spondylitis Metrology Index | 6 months
  Spinal mobility will assessed and scored by Bath Ankylosing Spondylitis Metrology Index (BASMI). There are five measurements including lateral lumbar flexion, tragus-to-wall distance, lumbar flexion (Modified Schober), maximal intermalleolar distance and cervical rotation according to the index. Each subscale is scored between 0 and 10. All points are then averaged to calculate total score. Higher values represent worse outcomes.
Bath Ankylosing Spondylitis Disease Activity Index | 6 months
  Bath Ankylosing Spondylitis Disease Activity Index which consists of 6 questions will be used to evaluate disease activity. BASDAI is a composite index, consisting of an assessment on a 10 cm horizontal visual analog scale of fatigue, axial pain, peripheral pain, enthesopathy and stiffness. Fifth and sixth questions are averaged. Addition to this score, other questions are averaged. Total score is between 0 and 10. Higher score represent worse outcome.
Lumbopelvic stabilization assessment | 6 months
  Lumbopelvic stabilization will be evaluated by a pressure biofeedback unit (Stabilizer Pressure Biofeedback Unit, Chattanooga Group Inc., Hixson, TN, USA). The participant will be positioned in crook lying position and the pressure cell will be placed under the lumbar spine and inflate to the baseline pressure of 40 mmHg. The participant will be instructed to perform abdominal hollowing without moving their spine or pelvis, and to hold the contraction for 10 seconds monitored by using a digital watch. The change in pressure during abdominal hollowing will be repeated three times and the mean of all the measurements will be recorded.
Disease-Related Functional Status | 6 months
  Bath Ankylosing Spondylitis Functional Index (BASFI) was used to assess the functional status. BASFI includes 10 items which eight of them related to physical limitations, and two of them inquiry about the coping strategies in daily life. Each item is scored between 0 and 10 (0: easy, 10: impossible) by the patient. The total score is calculated by summing all the items and dividing them to 10. Higher scores indicate a higher level of functional limitations.
Disease-Related Quality of Life | 6 months
  Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) will be used to evaluate the disease-related quality of life. It includes 18 yes/no questions. Each yes answer is scored as onepoint. ASQoL is a valid and reliable tool for both clinical purposes and scientific research. Higher scores indicate poorer quality of life.
Musculoskeletal Health Questionnaire | 6 months
  The Arthritis Research UK Musculoskeletal Health Questionnaire (MSK-HQ) is composed of 14 items which evaluate the holistic impact of different musculoskeletal diseases on a person's health over the last two weeks, regardless of the location of their musculoskeletal pain. These items consist of the severity of stiffness/pain (during the day and night), physical function (washing/dressing and walking), level of physical activity, symptom interference (with daily routine, work and social activities), needing help, trouble with sleeping, low energy/fatigue level, emotional well-being (mood and anxiety), understanding of treatment and diagnosis, confidence to self-management, independence and general impact of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: ADEM KÜÇÜK, Dr., Study Chair — Necmettin Erbakan University, Faculty of Medicine, Meram/KONYA/TURKEY
Locations (1):
- Yasemin Akkubak, Konya, Meram, Turkey (Türkiye)